CLINICAL TRIAL: NCT06491030
Title: The Use of a Novel Post-Operative Thoracolumosacral Orthosis for Prevention of Proximal Junctional Kyphosis After Adult Spinal Deformity Surgery
Brief Title: Post-Operative Thoracolumosacral Orthosis for PJK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Aspen Medical Products (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-2446
Record Dates: First submitted 2024-06-20; First posted 2024-07-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Proximal Junctional Kyphosis; Adult Spinal Deformity Surgery; Thoracolumbosacral Orthosis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Thoracolumosacral Orthosis (Experimental): Patients randomized to this arm will be fitted with an Aspen Medical Products "Align PJK™" TLSO brace. This is a 3-point, rigid hyperextension TLSO brace which is currently FDA approved under a 510k exemption but not commercially available. With this brace, the sternal pad height/width and belt component will be adjusted to optimize patient position and comfort. The brace will also be fitted with an external temperature sensing probe. Patients will be instructed to wear the brace at all times, including when in bed for 6-weeks post-operatively. At the 6-week visit patients will be asked to self-report compliance with the brace
  Interventions: Device: Align PJK™ TLSO brace
- No brace (Placebo Comparator): Patients in the control arm will be treated without a brace but will have no other differences in their post-operative treatment protocol. This will be considered "usual care" for the purposes of this study.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Align PJK™ TLSO brace — Patients will get randomized to receiving and wearing a back brace for 6 weeks postoperatively.
  Arms: Thoracolumosacral Orthosis
Other: Standard of Care — Patients will receive the standard of care postoperative instructions without a brace
  Arms: No brace

SUMMARY:
Proximal junctional kyphosis (PJK) is a common post-operative radiographic finding after surgery for adult spinal deformity (ASD) patients. Although the clinical relevance of isolated PJK is unclear, PJK can progress to symptomatic proximal junctional failures which requires a large revision surgery. Currently, post-operative bracing with a thoracolumbosacral orthosis (TLSO) is common practice after spinal deformity surgery, however the efficacy of this in preventing PJK is unknown. This multi-center randomized control trial identified 84 patients undergoing thoracolumbosacral fusion for ASD and plans to study the efficacy of a novel post-operative TLSO in preventing the development of PJK as defined by the proximal junctional angle on 6-month post-operative X-rays.

ELIGIBILITY:
Inclusion Criteria:

* 30-75-years-old
* Undergoing primary thoracolumbosacral fusion for ASD with an upper instrumented vertebrae (UIV) between T8-L2 and lower instrumented vertebrae (LIV) of S1 or the ilium.

Exclusion Criteria:

* Osteoporosis (defined as a T-score <-2.5 at the time of surgery)
* Body mass index (BMI) >35 kg/m2
* Revision fusions
* Fusions for trauma
* Those with a neuromuscular etiology for their deformity (i.e. Parkinson's disease, cerebral palsy, post-stroke, etc.)
* An underlying inflammatory arthropathy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of proximal junctional kyphosis development | This will be measured via scoliosis radiographs at the pre discharge, 6-week, and 6-month time points.
  As defined by a proximal junctional angle both ≥10° and 10°greater than pre-operative values.

SECONDARY OUTCOMES:
Change in patient reported outcome measures | 6 week and 6-month time points
  VAS leg pain, and VAS back pain (scale of 0-10). 0= no pain; 10=worst possible pain
Change in patient reported outcome measures | 6 week and 6-month time points
  Oswestry Disability Index (0-20% minimal disability; 21-40% moderate disability; 41-60% severe disability; 61-80 cripple, pain impinges on all aspects of life; 81-100% patients are bed bound)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Indiana Spine Group, Carmel, Indiana
  - University of Kansas, Overland Park, Kansas
  - Hospital for Special Surgery, New York, New York
  - University of Texas Health, Houston, Bellaire, Texas
  - Texas Back Institute, Dallas, Texas
  - Virgina Mason Franciscan Health, Seattle, Washington